CLINICAL TRIAL: NCT06095908
Title: The Effect of Ultrasound-Guided Bilateral Rectus Sheath Block Versus Wound Infiltration on Postoperative Pain in Gynecooncological Patients Undergoing Laparotomy With Midline Incision: Randomized Controlled Triple Blinding Study
Brief Title: The Effect of Bilateral Rectus Sheath Block Versus Wound Infiltration in Gynecooncological Patients
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Bulun Yediyıldız, Specialist Dr, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: DrLutfiKirdarANESTESIA
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
Keywords: postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 'rectus sheath block': Patients in Group I underwent postoperative USG-guided bilateral rectus sheath block at the T9-10 level with 20 ml of 0.25% bupivacaine (40 ml in total).
  Interventions: Drug: Bupivacain
- 'wound infiltration': Group II (control group), 20 ml of 0.25% bupivacaine was applied subcutaneously to each wound lip (40 ml in total).
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — Bupivacain administered with two different ways to the patients, postoperative pain recorded

SUMMARY:
Postoperative pain is a serious problem in gynecological oncology patients who underwent median vertical incision. The aim of our study is to compare ultrasound guided bilateral rectus sheath block and local anesthetic wound infiltration application in postoperative pain control.

DETAILED DESCRIPTION:
This single-center prospective,observational study was approved by Institutional Ethics Committee (Decision number: 2023/514/257/31, Date: 29/05/2023) and was performed in accordance with the Declaration of Helsinki.. Between June and September 2023, ultrasound guided bilateral rectus sheath block or local anesthesia administered to the patients in the gynecological oncology operating room of the University of Health Sciences Kartal Dr Lutfi Kırdar City Hospital at the end of the surgery. In the postoperative period, the pain level of the patients was recorded with the numerical rating scale at 2, 6, 12 and 24 hours by an anesthesiologist who was unaware of the application. The data were entered into the table by an anesthesiologist who did not know which application was performed. Thus, data were recorded using a randomized triple blinding method in which the patient, the researcher, and the recording staff were blinded.

All patients underwent preoperative evaluation one day before surgery and written informed consent was obtained for participation for the study. The procedure to be performed on the patients was planned in accordance with the randomization made by the statistician. The anesthesiologist who would perform the intervention participated in the study blindly to the drugs and groups. Patients in Group I underwent postoperative ultrasound-guided bilateral rectus sheath block at the T9-10 level with 20 ml of 0.25% bupivacaine (40 ml in total). For the patients in Group II (control group), 20 ml of 0.25% bupivacaine was applied subcutaneously to each wound lip (40 ml in total). At the end of the surgery, 100 mg tramadol iv and paracetamol 1mg/kg iv were administered to both groups as analgesics.

Pain, ranging from 0 (no pain) to 10 (worst imaginable), was queried by another anesthesiologist who was blind to the procedure. 2*1 non-steroidal anti-inflammatory was routinely administered as an analgesic in the ward, but the first application time was planned by questioning the patient's pain. Rescue analgesia with tramadol was administered if the patient ranged the pain >4 . Pain was measured at the 2nd, 6th, 12th and 24th hours postoperatively, and tramadol consumption was recorded.

ELIGIBILITY:
Inclusion Criteria:

* electively gynecooncological surgery patients with median incision
* ASA II-III,
* between 18-65 years

Exclusion Criteria:

* ASA IV and above
* over 65 - under 18 years of age
* previous laparotomy
* allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Between June and October 2023, 60 patients aged ASA II-III, 18-65 years old, who will undergo elective gynecooncological surgery with median incision will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluate patients' postoperative pain | postoperative 2,6,12,24 th hours
  The primary aim of this study is to evaluate and compare the postoperative analgesic effectiveness of bilateral rectus sheath block and wound infiltration in gyneco-oncological patients undergoing laparatomy with midline incision. Numeric rating scale (NRS) of 1-10 used for the assessment of postoperative pain.

SECONDARY OUTCOMES:
Evaluate patients' total analgesic consumption | postoperative 24 hours
  The secondary aim of the study was to evaluate the patients in terms of time to total amount of opioid analgesics (mg ) consumed in 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kırdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided